CLINICAL TRIAL: NCT00004419
Title: Study of Recombinant Human Insulin-Like Growth Factor I in Patients With Severe Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Masking: None | Purpose: Treatment
Other Study IDs: 199/13313; BIH-98-1060; BIH-E-147; BIH-FDR001126
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1999-06

CONDITIONS: Insulin Resistance; Hyperglycemia
Keywords: endocrine disorders; insulin resistance; rare disease
MeSH Terms: conditions — Insulin Resistance; Hyperglycemia; Endocrine System Diseases; Rare Diseases | interventions — Insulin-Like Growth Factor I

INTERVENTIONS:
Drug: insulin-like growth factor I

SUMMARY:
OBJECTIVES: I. Determine the efficacy and toxic effects of recombinant human insulin-like growth factor I (rhIGF-I) on carbohydrate tolerance, insulin action, insulin secretion, hyperandrogenism, and hyperlipidemia in patients with severe insulin resistance who have failed other therapies.

II. Determine the dose and time response of rhIGF-I on carbohydrate homeostasis and secondary abnormalities in this patient population.

III. Determine the effect of rhIGF-I on insulin clearance, the regulation of insulin-like growth factor binding protein 1, the regulation of sex hormone binding globulin, and hypothalamic pituitary gonadal axis in this patient population.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is an open label study. Patients receive the first dose of subcutaneous recombinant human insulin-like growth factor I (rhIGF-I) on day 7.

Patients receive rhIGF-I twice daily 15-30 minutes before breakfast and dinner, and are hospitalized for the first week of therapy. Patients return for an outpatient exam on day 19 of rhIGF-I therapy. Approximately 30 days into the therapy, patients are readmitted to the clinical center for repeat screening tests. Patients then receive maintenance therapy of rhIGF-I for up to 6-12 months. A washout period follows the maintenance therapy phase.

Patients are followed weekly, biweekly, or monthly depending on blood glucose response of patients off rhIGF-I therapy. Weekly phone contact with study coordinator is mandatory during this time.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Hematologically proven severe insulin resistance with or without diabetes
* Fasting insulin greater than 40 U/mL
* Post glucose insulin greater than 300 U/mL (unless overt diabetes mellitus is present)

--Prior/Concurrent Therapy--

Endocrine therapy: No concurrent oral hypoglycemic agents and/or insulin

Other: No concurrent birth control pills

--Patient Characteristics--

* Not pregnant
* Negative pregnancy test
* Effective barrier contraceptive method must be used by fertile patients
* Good health

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 1998-04; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Overall Officials: Alan C. Moses, Study Chair — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States